CLINICAL TRIAL: NCT01842178
Title: Randomized Prospective Study of Endometrial Injury in In Vitro Fertilization Cycles With Oocyte Donation
Brief Title: Endometrial Scratching in In Vitro Fertilization Cycles With Oocyte Donation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator retired from the project
Sponsor: Centro de Infertilidad y Reproducción Humana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRH-OLE:2013
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- scratching (Experimental): Patients will have an endometrial injury done on purpose, between 18-24 days prior to IVF cycle with a transfer catheter on the surgery outpatient department.
  Endometrial Injury
  * Done between 18-24 days prior to embryo transfer cycle.
  * Using transfer catheter.
  * Introduction of the same to the uterine fundus.
  * Systematic scrapping of the four uterine walls, lengthwise.
  * Performed by a skilled doctor.
  * Subsequent ultrasound control
  Interventions: Procedure: scratching
- scratching simulation (Placebo Comparator): Patients will come to control visit between day 18-24. A scratching simulation will be done.
  Interventions: Procedure: scratching

INTERVENTIONS:
Procedure: scratching — Endometrial Injury
  * Done between 18-24 days prior to embryo transfer cycle.
  * Using transfer catheter.
  * Introduction of the same to the uterine fundus.
  * Systematic scrapping of the four uterine walls, lengthwise.
  * Performed by a skilled doctor.
  * Subsequent ultrasound control.
  Other Names: endometrial enjury

SUMMARY:
This study is designed to evaluate the potential benefit in pregnancy rates produced by an endometrial scratching made in an IVF cycle prior to embryo transfer in patients with donated oocytes.

DETAILED DESCRIPTION:
This is a randomized, comparative, prospective, double Blind study.

The First stage of this study consists of revising the patients medical records to identify possible candidates. Patients indicated are randomized into two groups: experimental and control. They are followed up to 12 week of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Do IVF cycle with donor eggs
* Will adjust to protocol for the study.
* Have signed informed consent

Exclusion Criteria:

* Clinically significant systemic disease, hypothalamic or pituitary tumors
* ovarian, uterine or breast cancer
* hormonal abnormalities and / or medical , biochemistry, hematology pathology, which might interfere with gonadotropin treatment.
* known positivity for human immunodeficiency virus (HIV), hepatitis C or B virus (HCV / HBV) of the candidate or her partner.
* Uterine Factor(submucosal fibroids, intramural fibroids> 4 cm)
* Hydrosalpinx
* Patients receiving immune treatment
* Positive Diagnosis Thrombophilia
* preimplantation genetic diagnosis needed
* In case of using marital sperm are excluded the following patients:Altered male karyotype, Altered Meiosis in testicular biopsy, Altered FISH, sperm Fragmentation> 45%
* Pregnancy contraindication
* Known allergy to preparations containing estrogens or any of its excipients.
* Simultaneous participation in another clinical trial with medication.
* Do not want or can not adjust to study protocol.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
biochemical pregnancy | 14-16 days post-follicular punction
  Determination of human chorionic gonadotropin blood levels.

SECONDARY OUTCOMES:
Clinical pregnancy | 6 pregnancy weeks
  Ultrasound

OTHER OUTCOMES:
Evolutionary pregnancy | 12 weeks of pregnancy
  telephone patient contact
abortion | 6-12 week of pregnancy
  telephone contact of patients

CONTACTS AND LOCATIONS:
Overall Officials: miguel angel checa, MD, Study Director — Centro de Infertilidad y Reproducción Humana
Locations (1):
- Centro de Infertilidad y Reproducción Humana, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No